CLINICAL TRIAL: NCT05962606
Title: An Exploratory, Multi-Centre, Interventional, Prospective, Randomised, Double-Blind, Placebo-Controlled Clinical Trial to Assess the Safety and Efficacy of AON-D21 in Patients With Severe Community-Acquired Pneumonia.
Brief Title: Safety and Efficacy of AON-D21 in Severe Community-Acquired Pneumonia.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aptarion Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-D21-C300
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia; Community-acquired; Severe; Bacterial; Viral
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Multi-center, interventional, randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AON-D21 plus Standard of Care (Experimental): Sterile liquid formulation of AON-D21 in 4% mannitol + 0.05% EDTA in glass vials. It will be administered intravenously, for up to 10 days plus Standard of Care therapy for severe community-acquired pneumonia as per local guidelines.
  Interventions: Drug: AON-D21
- Placebo plus Standard of Care (Placebo Comparator): Sterile liquid formulation of 5% glucose solution in matched glass vials with a 1.5 mL fill volume. It will be administered intravenously, for up to 10 days plus Standard of Care therapy for severe community-acquired pneumonia as per local guidelines.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AON-D21 — AON-D21 is a Pegylated L-configured aptamer that binds and thereby neutralizes the complement component C5a from activating both C5a receptors.
  Arms: AON-D21 plus Standard of Care
Drug: Placebo — Sterile liquid formulation of 5% glucose solution in matched glass vials with a 1.5 mL fill volume.
  Arms: Placebo plus Standard of Care

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy of AON-D21 versus placebo, both on top of standard of care, in patients with severe community acquired pneumonia admitted to ICU (or similar unit). The main questions to answer are:

* The safety and tolerability of AON-D21 vs placebo.
* The efficacy of AON-D21vs placebo.
* The pharmacokinetics of AON-D21.
* The pharmacodynamics of AON D21.
* To identify biomarkers for patient stratification and analyses in future trials.

DETAILED DESCRIPTION:
This clinical trial will enroll 100 participants, randomized 2:1 (AON-D21:placebo).

Participants diagnosed with severe community-acquired pneumonia of bacterial or viral origin requiring admission to an intensive care unit or similar setting, will receive either AON-D21 or placebo intravenous infusions for up to 10 days.

In addition, participants will receive standard of care as per local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Community-acquired pneumonia, confirmed or suspected of bacterial or viral origin.
* Admitted to an ICU (or similar unit).
* Requiring respiratory support by HFO ≥ 30 L/min with FiO2 ≥ 30% or NIV or IMV or ECMO.
* CRP ≥ 50 mg/L.
* PaO2/FiO2 ratio ≤ 150 mmHg.
* Treatment initiation no more than 48 h after initiation of respiratory support (HFO ≥ 30 L/min with FiO2 ≥ 30%, NIV, IMV or ECMO).
* Written informed consent.
* Age ≥ 18 years to ≤ 85 years.
* Body mass index ≥ 17.5 kg/m² and ≤ 40 kg/m².
* For female participants of childbearing potential, agreement to use dual methods of contraception until Day 60.
* For male participants with female partners of childbearing potential, agreement to use barrier method of contraception until Day 60 and to refrain from donating sperm during the study and for 3 months after the last infusion.

Exclusion Criteria:

* Refractory septic shock.
* Not expected to survive 72 hours.
* Hospital-acquired or ventilator-associated pneumonia or known or suspected pneumonia due to aspiration or other physical injury or trauma or tuberculosis.
* Known or suspected hypersensitivity to AON-D21 or any components of the formulation used (e.g., PEG, mannitol or EDTA) or a history of clinically relevant allergy requiring continuous treatment, or of anaphylaxis.
* Known fibrotic lung disease, bronchiectasis or any other known severe chronic respiratory disease.
* Active malignant disease.
* Factors other than a pathogen suspected or confirmed to be causative for the respiratory insufficiency.
* Hepatocellular injury defined by an ALT or AST value ≥ 3 times the ULN. Known acute or chronic liver disease with Child-Pugh C (See Appendix 13.6.2).
* Any medical disease or condition that, in the opinion of the investigator(s), compromises the participant's safety or compromises the interpretation of the results.
* Receiving chronic immunosuppressive therapy in relevant doses.
* Known immunodeficiency disease/condition.
* Nursing and pregnant women (defined as the state after conception until the termination of gestation, screened in all women of child-bearing potential with a chorionic gonadotrophin (hCG) blood test (local laboratory).
* Current or recent participation in an investigational trial.
* Systemic treatment with any complement inhibitor.
* Known complement deficiency.
* Unlikely to remain at the investigational site beyond 96 h.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events. | 28 days.
  To evaluate the safety and tolerability of AON-D21 versus placebo, including the frequency, severity, and relatedness to study drug of serious and non-serious treatment-emergent adverse events (TEAEs) until Day 28.

SECONDARY OUTCOMES:
Efficacy-no longer requiring respiratory support. | 28 days.
  Comparing AON-D21 vs placebo on time to no longer requiring respiratory support (defined as high-flow oxygen (HFO) ≥ 30 L/min with FiO2 ≥ 30%), non-invasive mechanical ventilation (NIV), invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) within 28 days.
Efficacy-no longer requiring any organ support. | 28 days.
  Comparing AON-D21 vs placebo on time no longer requiring any organ support within 28 days.
Efficacy-time to improvement. | 28 days.
  Comparing AON-D21 vs placebo on time to improvement (defined as a de-escalation in respiratory support) within 28 days.
Efficacy-mean change in SaO2/FiO2 ratio. | 7 days.
  Comparing AON-D21 vs placebo on mean change in SaO2/FiO2 ratio from Day 1 (Baseline) to Day 7.
Efficacy-organ support-free days. | 28 days.
  Comparing AON-D21 vs placebo on organ support-free days until Day 28.
Efficacy-invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO)-free days. | 28 days.
  Comparing AON-D21 vs placebo on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO)-free days until Day 28.
Efficacy-respiratory support-free days. | 28 days.
  Comparing AON-D21 vs placebo on respiratory support-free days until Day 28.
Efficacy-all-cause mortality. | 28 days.
  Comparing AON-D21 vs placebo on all-cause mortality up to Day 28.
Efficacy-all-cause mortality. | 60 days.
  Comparing AON-D21 vs placebo on all-cause mortality up to Day 60.
AUC of AON-D21. | 10 days.
  Area under the concentration-time curve (AUC) over the dosing interval at steady state (AUC0-tau).
Cmax of AON-D21. | 10 days.
  Maximum concentration at steady state (Cmax)
Cav of AON-D21. | 10 days.
  Average drug concentration at steady state (Cav).
Ctrough of AON-D21. | 10 days.
  Trough concentrations (Ctrough).
Tmax of AON-D21. | 10 days.
  Time of maximum concentration at steady state (Tmax).
Half-life of AON-D21. | 12 days.
  Terminal half-life at steady state (t1/2).
Accumulation of AON-D21. | 10 days.
  Accumulation ratio for Cmax.
Clearance of AON-D21. | 12 days.
  Clearance (CL).
Volume of distribution of AON-D21. | 12 days.
  Volume of distribution (Vz).
C5a inhibition with AON-D21. | 12 days.
  To determine the C5a inhibition capacity of AON-D21 by measuring active C5a in blood using a cell-based assay.
Procalcitonin's measurement. | 12 days.
  Evolution of procalcitonin over time.
Ferritin's measurement. | 12 days.
  Evolution of ferritin over time.
IL-6's measurement. | 12 days.
  Evolution of IL-6 over time.
C5a's measurement | 12 days.
  Evolution of C5a over time.
sC5b-9's measurement. | 12 days.
  Evolution of sC5b-9 over time.
Neutrophil elastase's measurement. | 12 days.
  Evolution of neutrophil elastase over time.
D-dimer's measurement. | 12 days.
  Evolution of D-dimer over time.
Pro-Adrenomedullin's measurement. | 12 days.
  Evolution of Pro-Adrenomedullin over time.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Witzenrath, MD, Principal Investigator — Critical Care Medicine. Charité Universitätsmedizin Berlin
Locations (27):
- University of Alabama at Birmingham Heersink School of Medicine, Birmingham, Alabama, United States
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Clinique Saint Pierre, Ottignies
- France (9):
  - Centre Hospitalier Argenteuil, Argenteuil
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - CHU Dupuytren, Limoges
  - Centre Hospitalier de Melun, Melun
  - Hotel Dieu - CHU Nantes, Nantes
  - Assistance Publique-Hopitaux de Paris (AP-HP), Paris
  - Nouvel Hôpital Civil, Strasbourg
  - CHRU de Tours Hôpital Bretonneau, Tours
  - Hôpital Nord Franche Comté, Trévenans
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Cologne-Merheim Hospital Lung Clinic, Cologne
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Doctor Josep Trueta, Girona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (8):
  - University Hospital Bristol and Weston NHS, Bristol
  - University Hospital of Wales, Cardiff
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - University College London, London
  - University Hospitals Plymouth NHS Trust, Derriford Hospital, Plymouth
  - Royal Berkshire Foundation Trust, Reading
  - Mid Yokshire Teaching NHS Trust, Wakefield
  - York Hospital, York

IPD SHARING:
Plan to Share IPD: No